CLINICAL TRIAL: NCT03267875
Title: A Laboratory Scan of Patients With Aortic Aneurysms to IgG4 Levels in the Blood
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, yair levy, Professor, Meir Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Aneurysm-IgG4
Record Dates: First submitted 2017-08-29; First posted 2017-08-30 (Actual); Last update posted 2017-11-09 (Actual); Status verified 2017-08

CONDITIONS: IgG4-related Disease; Aortic Aneurysm
MeSH Terms: conditions — Immunoglobulin G4-Related Disease; Aortic Aneurysm | interventions — Hematologic Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Patients after aneurysm in the aorta, Men and women aged 18-100 (not including special populations), who are able to read understand and sign a written consent to participate in the research
  Interventions: Procedure: Blood Test

INTERVENTIONS:
Procedure: Blood Test — draw out 2 blood tubes from a patient

SUMMARY:
IgG4 Related Disease is a multi-systemic fibroenophilic disease that includes a basket of recently discovered medical conditions.

The properties that bind them are: lesions similar to tumors in the mixed organs, lymphoplasms filtrate enriched with plasma IgG4 positive cells, storiform fibrosis, and often, but not always, a high level of IgG4 in the serum.

This disease has been on the rise for the past two decades and since its recognition in 2001 there has been impressive progress in understanding its various manifestations, so that today almost every body system can be involved.

One of the conditions associated with this disease is oritis / periortitis and aneurysms

DETAILED DESCRIPTION:
IgG4 Related Disease is a multi-systemic fibroenophilic disease that includes a basket of recently discovered medical conditions.

The properties that bind them are: lesions similar to tumors in the mixed organs, lymphoplasms filtrate enriched with plasma IgG4 positive cells, storiform fibrosis, and often, but not always, a high level of IgG4 in the serum.

This disease has been on the rise for the past two decades and since its recognition in 2001 there has been impressive progress in understanding its various manifestations, so that today almost every body system can be involved.

One of the conditions associated with this disease is oritis / periortitis and aneurysms

It is common to divide the aortic aneurysms according to the following etiologies:

1. Inflammatory-Aortic Aneurisms (IAA) The internal division in this category is whether IgG4RD is related / not related.
2. Atherosclerotic infrastructure.

Differences between the etiologies: IAA - greater thickness of the wall, fibrosis and adhesion to nearby retroperitone structures. Also, younger age and non-specific symptoms. In addition, the laboratory findings are usually white counts and increased CRP.

In this context, the investigators will examine the level of IgG4 in the blood of a population of patients with aortic aneurysms and try to understand the proportion of patients whose IgG4 level is higher than normal and their aneurysm can be attributed to IgG4 Related Disease.

the investigator chose the blood IgG4 level because it is the most important diagnostic variable for the disease (it is customary to place the incision point at > 135mg / dL).

ELIGIBILITY:
Inclusion Criteria:

* Patients after aneurysm in the aorta
* Men and women aged 18-100 (not including special populations)
* Those who are able to read understand and sign a written consent to participate in the research

Exclusion Criteria:

* Any patient who does not meet the inclusion criteria

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — male and female
Enrollment: 300 (Estimated)
Dates: Start 2017-11-08 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
IgG4 Level | 1 year
  count IgG4 Level to figure if its IgG4-related disease

CONTACTS AND LOCATIONS:
Overall Officials: Yael Eizikovits, B.A, Study Chair — Meir Medical Center
Locations (1):
- Yael Eizikovits, Kfar Saba, Israel

IPD SHARING:
Plan to Share IPD: Undecided